# 临床研究知情同意书

### 尊敬的受试者:

您将被邀请参加一项由福建医科大学附属第一医院张文明主任医师(项目负责人)(电话号码: 13950391800)主持的研究,研究项目名称:利福平联合抗生素治疗葡萄球菌假体周围感染的疗效与并发症——一项多中心、随机对照试验。

您参加本项研究是自愿的,本知情同意书提供给您一些信息以帮助您决定是否参加此项临床研究。本研究已通过福建医科大学附属第一医院伦理委员会审查同意,伦理委员会办公室电话 0591-87981029。如果您同意加入此项研究,请您仔细阅读,如有任何疑问请向负责该项研究的研究者提出。

#### 一、研究目的:

假体周围感染(PJI)是关节置换手术后常见且严重的并发症,给患者带来了巨大的痛苦和治疗挑战。 PJI 不仅会延长住院时间,还可能导致手术失败和严重的健康后果。因此,如何有效控制和治疗这种感染成为临床医生关注的重点。在这一过程中,抗生素的使用显得尤为重要,它们是对抗感染的主要武器。

目前,对于 PJI 术后的抗生素治疗方案中是否应添加利福平,以提高感染控制效果,医疗界仍然存在较大分歧。一些研究认为利福平能够增强抗生素的效果,帮助更好地控制感染;而另一些研究则对其具体效果提出质疑,认为需要更多的证据来支持这一做法。由于这些争议,临床实践中对利福平的使用缺乏统一的标准。

为了解决这一问题,我们计划开展一项多中心随机对照临床试验,专门研究联合利福平治疗对 PJI 感染控制的影响。这项研究将汇集多家医院的参与,确保样本的多样性和结果的可靠性。通过严谨的设计和科学的数据分析,我们希望能够明确利福平在 PJI 治疗中的具体作用。

我们的目标是为优化临床抗生素治疗方案提供有力的证据支持,从而帮助医生们在面对这种复杂感染时做出更好的决策。这不仅有助于改善患者的预后,也为今后的临床治疗提供了重要的参考依据。

#### 二、研究过程和方法:

如果您同意参与这项研究,我们将为每位受试者分配一个编号,并建立详细的研究档案。本研究将筛选出病原菌为革兰氏阳性菌的 PJI 患者,在经过手术治疗后,随机分为利福平联合抗生素治疗组和常规抗生素治疗组。在研究期间,患者需要定期复诊,医生将评估感染复发率、炎症指标、假体功能恢复及药物副作用等情况。所有相关数据将被统一记录,并在随访结束后进行分析,以比较两组在疗效和安全性方面的差异。通过这项研究,我们期望明确利福平联合治疗的效果,从而为 PJI 抗生素治疗方案的优化提供重要依据。

在接受抗生素治疗后的第 2 周、1 个月、3 个月、6 个月、12 个月、18 个月和 24 个月时,您需要按时回到医院进行复诊,并如实向医生反馈您的病情变化。医生将收集您的病史,并进行常规复查和体检,包括血常规、CRP、ESR、肝肾功能等理化检查。在治疗后的第 24 个月,即出院后 2 年时,研究将结束,您需要再次回到医院进行复诊。医生将询问并记录您的病情变化,并进行体格检查,为您安排必要的血常规、CRP、ESR、肝肾功能等理化检查。

## 三、研究可能的受益:

参与在本研究您可能不会直接受益,但也有可能因为您的参与,您和社会都会从中获益。这些潜在的 益处包括您的病情可能得到改善,同时本研究可能为 PJI 抗生素治疗方案提供新的认知,从而帮助类似病情 的其他患者。

## 四、研究风险与不适:

## 1、服用抗生素所带来的风险:

- 1) **为所有入组患者购买保险**,在研究过程中,使用抗生素可能会带来一些副作用。常见的风险包括过敏反应、急性肾功能不全、间质性肾炎等肾功能损害,以及肝功能损害、黄疸、多种血细胞减少、中枢神经系统、消化系统、生殖系统和心血管系统的损害。如果您出现上述任何不良反应,医生将立即停止药物使用,并采取适当的治疗措施,以确保您的健康和安全,并视实际情况由保险公司理赔。
- 2) 抗生素可能与其他药物发生相互作用,从而引发副作用。为了您的安全,请在参与本研究前告知医生您正在服用的所有药物,包括处方药、中草药、非处方药、维生素,以及您是否正在接受其他自然疗法或饮用含酒精的饮品等。
  - 3) 耐药菌: 抗生素的使用可能会导致病原微生物产生耐药性,从而引发耐药菌的出现。

## 2、可选择的其他诊疗方法:

您有权拒绝参加该研究,或者咨询您的主治医生关于其他常规治疗方法,包括但不限于喹诺酮类抗生素治疗(例如:环丙沙星、左氧氟沙星、莫西沙星等)。同时,我们也会尽心为您提供最好的诊疗服务,确保您的健康和安全。

## 五、隐私问题: (过程中的隐私保护和结果发表的隐私保护)

如果您决定参加本项研究,您参加试验及在试验中的个人资料均属保密。对于您来说,所有的信息将是保密的。所有的研究成员和研究申办方都被要求对您的身份保密。您的档案将保存在福建医科大学附属第一医院科研处档案柜中,仅供研究人员查阅。为确保研究按照规定进行,必要时,政府管理部门或伦理审查委员会的成员按规定可以在研究单位查阅您的个人资料。该项研究结果发表时,也会对您的身份信息进行保密。

#### 六、费用

如果您选择参与本研究项目,手术期间的诊疗费用以及术后随访的理化检查费用将与您正常接受治疗时产生的费用相同。这些费用是标准医疗过程中的一部分,并不因您参与研究而增加额外费用。在您参与本研究项目的期间,我们将为您提供利福平药物,且不收取任何费用。以下是您的治疗方案详述:

您将被纳入联合抗生素治疗组。在此治疗组中, 您将接受以下药物治疗:

- 1、常规抗生素治疗,作为基础治疗方案。
- 2、利福平治疗,作为研究干预措施的一部分,如果您被分配至利福平联合抗生素治疗组,您将在常规 抗生素治疗基础之上,额外还需口服利福平,治疗至满三个月。

利福平的市场单价为 22.93 元人民币,药品规格为 0.15 克×100 粒。作为本研究的一部分,您在研究期间使用该药物将不会承担任何费用。

# 七、补偿

1) 如果在临床试验中出现不良事件,研究医师将及时采取积极措施进行治疗。

### 八、自由退出:

作为受试者,您可随时了解与本研究有关的信息资料和研究进展,自愿决定(继续)参加还是不(继续)参加。参加后,无论是否发生伤害,您可以选择在任何时候通知研究者要求退出研究,您的数据将不纳入研究结果,您的任何医疗待遇与权益不会因此而受到影响。在试验过程中,若会对您造成严重的伤害,研究者也将会中止研究的进行。

但在参加研究期间,请您提供有关自身病史和当前身体状况的真实情况;告诉研究医生自己在本次研究期间所出现的任何不适;不得服用受限制的药物、食物等;告诉研究医生自己在最近是否曾参与其他研究,或目前正参与其他研究。如果因为您没有遵守研究计划,或者发生了与研究相关的损伤或者有任何其

它原因,研究医师可以终止您继续参与本项研究。

# 九、联系方式:

如果您有与本研究有关的问题,或您在研究过程中发生了任何不适与损伤,或有关于本项研究参加者 权益方面的问题,您可以与方心俞医生联系,电话 18084768503。

# 十、知情同意签字:

我已经阅读了本知情同意书,并且我的医生 (签字)已经将此次临床试验的目的、内容、风险和受益情况向我作了详细的解释说明,对我询问的所有问题也给予了解答,我对此项临床研究已经了解,我自愿参加本项研究。

| 受试者签名: | | | | 研究者签字: |
|--------------|-------|-------|------------|--------------|
| 联系手机号: | | | | 联系手机号: |
| 日期: | 年 | _月 | _日 | 日期:年月日 |
| (如果受试者 | 不识字时尚 | 需见证人签 | 名,如果受试者无行为 | 7能力时则需代理人同意) |
| 法定代理人/见证人签名: | | | | |
| 与受试者的关系: | | | | |
| 日期: | _年 | 月 | 日 | |